CLINICAL TRIAL: NCT01277042
Title: Immunogenicity and Safety Study of GSK Biologicals' HPV Vaccine (GSK 580299) in Healthy Adult Chinese Female Subjects
Brief Title: Study to Assess Immune Responses and Safety of the GSK-580299 Vaccine in Healthy Women (26 to 45 Years)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 114590
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-08

CONDITIONS: Infections, Papillomavirus
Keywords: Safety; HPV vaccine; Immune response; Human papillomavirus; China
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Cervarix Group (Experimental): Subjects received a 3-dose vaccination course of the Cervarix™ vaccine administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: GSK580299 (CervarixTM)
- Engerix Group (Active Comparator): Subjects received a 3-dose vaccination course of the Engerix™-B vaccine administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: Engerix-BTM

INTERVENTIONS:
Biological: GSK580299 (CervarixTM) — 3-dose schedule intramuscularly vaccination (Months 0, 1 and 6)
  Arms: Cervarix Group
Biological: Engerix-BTM — 3-dose schedule intramuscularly vaccination (Months 0, 1 and 6)
  Arms: Engerix Group

SUMMARY:
This study is designed to evaluate the immunogenicity and safety of GSK Biologicals' human papillomavirus (HPV) vaccine in adult female subjects aged 26-45 years. One group of subjects will receive the HPV vaccine and the other group will receive an active control (GSK Biologicals' hepatitis B vaccine). Immunogenicity data of the HPV group will be compared with those from the HPV group included in the NCT00779766 study (aged 18-25 years).

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol Amendment 1, December 2010, leading to:

* The removal of 3 outcome measures
* The update of 1 outcome measure

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to study enrolment.
* Healthy adult females from Chinese origin and residing in China between and including 26 and 45 years of age at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* Healthy subjects as established by medical history and history-directed clinical examination before entering into the study.
* Subjects must not be pregnant. Absence of pregnancy will be verified with a urine pregnancy test before each vaccination.

Subjects must be of non-childbearing potential, i.e., have a current tubal ligation, hysterectomy, ovariectomy, be one year post-menopausal, or if of childbearing potential, they must be abstinent or have practiced adequate contraception for 30 days prior to vaccination, have a negative pregnancy test on the day of vaccination and agree to continue such precautions during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after the first dose of vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* A subject planning to become pregnant, likely to become pregnant or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Pregnant or breastfeeding subjects must be at least three months post-pregnancy and not breastfeeding to enter the study.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the protocol during the study period.
* Previous administration of 3-O-desacyl-4'-monophosphoryl lipid A or AS04 adjuvant.
* Previous vaccination against hepatitis B or planned administration of any hepatitis B vaccine other than that foreseen by the study protocol during the study period.
* History of hepatitis B infection.
* Known exposure to hepatitis B within the previous 6 weeks.
* History of chronic condition(s) requiring treatment such as cancer or autoimmune disease.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the vaccine (e.g. aluminium).
* Hypersensitivity to latex.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 26 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1212 (Actual)
Dates: Start 2011-02-17; Primary Completion 2011-09-26 (Actual); Study Completion 2012-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Jintan, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Zhu F, Li J, Hu Y, Zhang X, Yang X, Zhao H, Wang J, Yang J, Xia G, Dai Q, Tang H, Suryakiran P, Datta SK, Descamps D, Bi D, Struyf F. Immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine in healthy Chinese girls and women aged 9 to 45 years. Hum Vaccin Immunother. 2014;10(7):1795-806. doi: 10.4161/hv.28702. PMID 25424785
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114590 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114590 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114590 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114590 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114590 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114590 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised a Primary Vaccination Phase from Day 0 to Month 7, followed by a Long-Term Safety Follow-up Phase, up to Month 12.
Period: Overall Study
Arm/Group | Cervarix Group | Engerix Group
Started | 606 | 606
Completed | 598 | 601
Not Completed | 8 | 5
Not completed — Adverse Event | 4 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Engerix Group | Total
Number analyzed (Participants) | 606 | 606 | 1212
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.8 (4.92) | 35.6 (5.06) | 35.7 (4.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 606 | 606 | 1212
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects Against Human Papillomavirus-16 (HPV-16) and HPV-18
Description: A seroconverted subject was defined as a subject seronegative at baseline whose concentration for anti-HPV-16/18 antibodies, as measured by Enzyme-linked Immunosorbent assay (ELISA) , was higher than or equal to (≥) cut-off value. A seronegative subject was defined as a subject whose antibody concentration was below (<) cut-off value. Cut-off values were 8 ELISA units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: One month after third vaccination (Month 7)
Population: The analysis was based on the according-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 365 | 401
Participants
  HPV-16: number analyzed (Participants) | 345 | 344
  HPV-16 | 345 | 67
  HPV-18 | 363 | 135

2. Secondary Outcome: Number of Subjects Seropositive Against HPV-16 and HPV-18
Description: A seropositive subject was defined as a subject whose anti-HPV-16/18 antibody concentration, as measured by ELISA, was higher than or equal to (≥) cut-off value. Cut-off values were 8 ELISA units per milliliter (EL.U/mL) for anti-HPV-16 antibodies, and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: Before vaccination (Month 0) and one month after third vaccination (Month 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 596 | 601
Participants
  HPV-16, Day 0 | 251 | 257
  HPV-16, Month 7 | 596 | 322
  HPV-18, Day 0 | 231 | 200
  HPV-18, Month 7 | 594 | 312

3. Secondary Outcome: Concentrations for Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: Concentrations are given as geometric mean titers (GMTs), expressed in ELISA units per milliliter (EL.U/mL). Cut-off values were 8 EL.U/mL for anti-HPV-16 antibodies, and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: Before vaccination (Month 0) and one month after third vaccination (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 596 | 601
EL.U/mL
  HPV-16, Day 0 | 9.7 [8.8 to 10.6] | 9.3 [8.5 to 10.2]
  HPV-16, Month 7 | 6439.8 [6039.8 to 6866.3] | 12.1 [11.0 to 13.4]
  HPV-18, Day 0 | 6.4 [6.0 to 6.9] | 6.0 [5.6 to 6.5]
  HPV-18, Month 7 | 3563.3 [3310.0 to 3836.0] | 8.7 [8.0 to 9.5]

4. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Grade 3 redness and swelling were redness and swelling above 50 millimeters (mm) and grade 3 pain was defined as pain that prevented normal activity. Any was defined as the incidence of a symptom regardless of intensity grade.
Time Frame: During the 7 days (Days 0 - 6) after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented and symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 604 | 606
Participants
  Any pain | 470 | 296
  Grade 3 pain | 36 | 5
  Any redness | 156 | 88
  Grade 3 redness | 2 | 1
  Any swelling | 146 | 58
  Grade 3 swelling | 11 | 1

5. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited symptoms were arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, urticaria and temperature [axillary temperature above (>)37 degrees Celsius(°C)].Grade 3 temperature= temperature >39°C. Grade 3 utricaria= distributed on at least 4 body areas. Grade 3 symptom=prevented normal activity. Gastrointestinal symptoms=nausea, vomiting, diarrhoea and/or abdominal pain. Arthralgia (joint pain): in joints distal from injection site. Any=incidence of a symptom regardless of intensity grade or relationship to vaccination. Related = incidence of a symptom assessed by investigator as related to vaccination.
Time Frame: During the 7 days (Days 0 - 6) after any vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 604 | 606
Participants
  Any arthralgia | 19 | 14
  Grade 3 arthralgia | 0 | 0
  Related arthralgia | 17 | 12
  Any fatigue | 100 | 68
  Grade 3 fatigue | 1 | 1
  Related fatigue | 93 | 59
  Any gastrointestinal symptoms | 33 | 24
  Grade 3 gastrointestinal symptoms | 1 | 0
  Related gastrointestinal symptoms | 24 | 11
  Any headache | 71 | 46
  Grade 3 headache | 4 | 0
  Related headache | 64 | 38
  Any myalgia | 69 | 42
  Grade 3 myalgia | 1 | 0
  Related myalgia | 66 | 39
  Any rash | 2 | 1
  Grade 3 rash | 0 | 0
  Related rash | 1 | 1
  Temperature >37.0°C | 28 | 24
  Temperature >39.0°C | 0 | 0
  Related temperature | 15 | 13
  Any urticaria | 4 | 1
  Grade 3 urticaria | 2 | 0
  Related urticaria | 3 | 1

6. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination, grade 3 was a SAE that prevented normal activities, and related was defined as a SAE assessed by the investigator to be causally related to the study vaccination. and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Throughout the study (from Month 0 up to Month 12)
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 606 | 606
Participants
  Any SAE(s) | 3 | 3
  Grade 3 SAE(s) | 2 | 0
  Related SAE(s) | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: Within 30 days (Days 0 - 29) after any vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 606 | 606
Participants
  Any AE(s) | 32 | 36
  Grade 3 AE(s) | 2 | 2
  Related AE(s) | 0 | 1

8. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions (MSCs) Including Potential Immune Mediated Diseases (pIMDs)
Description: MSCs were AEs prompting emergency room or physician visits that were not related to common diseases (upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury), or not related to routine visits for physical examination or vaccination. It also included SAEs not related to common diseases. MSCs included pIMDs, a subset of MSCs that included autoimmune diseases and other inflammatory and/or neurological disorders of interest which might or might not have had an autoimmune etiology.
Time Frame: Throughout the study (from Month 0 up to Month 12)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Engerix Group
Number analyzed (Participants) | 606 | 606
Participants | 5 | 7

9. Secondary Outcome: Number of Subjects With Outcome of Pregnancies
Description: The sole pregnancy outcome reported was elective termination with no apparent congenital anomaly.
Time Frame: Throughout the study (from Month 0 up to Month 12)
Population: The analysis was performed on Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented, solely on subjects with outcome of pregnancies.
Measure: Count of Participants; unit: Participants
Groups:
- Engerix-B Group: Subjects received a 3-dose vaccination course of the Engerix™-B vaccine administered intramuscularly in the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
Arm/Group | Cervarix Group | Engerix-B Group
Number analyzed (Participants) | 4 | 1
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from Month 0 up to Month 12. Systematically assessed frequent adverse events were assessed during 7 days (Days 0-6) post vaccination period.
Description: For the systematically assessed other (non-serious) adverse events the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | Cervarix Group | Engerix Group
Serious Adverse Events (participants affected / at risk) | 3/606 | 3/606
Other Adverse Events (participants affected / at risk) | 490/606 | 318/606
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=606) | Engerix Group (N=606)
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Gastroenteritis shigella (Infections and infestations) | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=606) | Engerix Group (N=606)
Pain (General disorders) | 470 | 296
Redness (General disorders) | 156 | 88
Swelling (General disorders) | 146 | 58
Fatigue (General disorders) | 100 | 68
Gastrointestinal (General disorders) | 33 | 24
Headache (General disorders) | 71 | 46
Myalgia (General disorders) | 69 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.